CLINICAL TRIAL: NCT01786161
Title: Prospective Evaluation of a Vancomycin Nomogram With a Continuous Infusion of Vancomycin for Surgical ICU Patients
Acronym: CIV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hsin Jung Lin, PharmD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 002617
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: MRSA - Methicillin Resistant Staphylococcus Aureus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin with continuous infusion (Experimental): 24 hours continuous infusion
  Interventions: Drug: Vancomycin continuous infusion
- Vancomycin with intermittent dose interval (Active Comparator): infusion rate 1000mg/hr
  Interventions: Drug: Vancomycin intermittent dosing interval

INTERVENTIONS:
Drug: Vancomycin continuous infusion — Vancomycin 24 hour intravenous continuous infusion
  Arms: Vancomycin with continuous infusion
Drug: Vancomycin intermittent dosing interval — Vancomycin intravenous infusion at rate 1000mg/hr
  Arms: Vancomycin with intermittent dose interval

SUMMARY:
Vancomycin is an essential antimicrobial which is frequently used in the ICU for suspected methicillin-resistant Staphylococcus aureus (MRSA) infection. Therefore, it is vital to optimize the dosing of vancomycin for this critically ill population. The most efficacious method of administering vancomycin is debated in the literature. Since vancomycin is associated with slow bactericidal activity, it is important to closely monitor serum concentrations so as to achieve early target serum concentration, particularly when treating aggressive S. aureus infections. One study has shown that vancomycin infused continuously may enable faster and more consistent achievement of a therapeutic serum concentration when compared to intermittent infusion. A faster achievement in the goal serum vancomycin concentration would be a protective factor for intensive care unit mortality in patients with MRSA infection.

Currently in the surgical ICU (SICU) of our institute, vancomycin is administered based on a vancomycin dosing nomogram. Less than fifty percent of the ICU patients following this nomogram achieved target vancomycin concentration of 15 after 24 hours. To better achieve target vancomycin concentration in 24 hours, we developed a new vancomycin dosing nomogram with a continuous infusion. The aim is to determine which of the two dosing nomogram is more efficient and safer for SICU patients.

DETAILED DESCRIPTION:
Early administration of effective antibiotics is the cornerstone of management in septic patients; however, altered pharmacokinetics in critically ill patients has lead to subtherapeutic antibiotic exposure with standard antibiotic dosing and administration. This is further evidenced by low therapeutic target achievement with our intermittent vancomycin dosing nomogram. Administering vancomycin by continuous infusions may lead to achieving a therapeutic concentration and AUC24 more quickly than the administration by intermittent infusions as well as provide a more consistent concentration throughout the dosing period. Therefore, a new vancomycin continuous infusion nomogram was developed to increase the achievement of a goal vancomycin concentration within 24 hours.

We hypothesized that vancomycin administered as continuous infusion would achieve the therapeutic target sooner and more consistently than when administered as an intermittent infusion in critically ill surgical patients. The aims of this study were to determine the dosing differences between continuous (CIV) and intermittent (IIV) dosing in critically ill surgical intensive care unit (SICU) patients with preserved renal function and whether calculated Cockcroft-Gault Creatinine Clearance (CG CrCL) or measured creatinine clearance (CrCL) is a better predictor of vancomycin clearance.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female > 18 years of age admitted to Surgical ICUs with suspected infection
* Calculated creatinine clearance > 60ml/min

Exclusion Criteria:

* Age < 18 years
* Allergic to vancomycin
* Calculated creatinine clearance < 60ml/min
* Pregnant
* Vancomycin administration more than 8 hour and less than 24 hour prior to study enrollment
* Anticipated vancomycin treatment less than 2 days for surgical prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin Lin, PharmD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin With Continuous Infusion: continuous 24 hours intravenous infusion
  Vancomycin continuous infusion: Vancomycin 24 hour intravenous continuous infusion
Period: Overall Study
Arm/Group | Vancomycin With Continuous Infusion | Vancomycin With Intermittent Dose Interval
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vancomycin Continous Infusion: Vancomycin continuous infusion: Vancomycin 24 hour intravenous continuous infusion infusion rate 1000mg/hr
- Intermittent Infusion: infusion rate 1000mg/hr
  Vancomycin intermittent dosing interval: Vancomycin intravenous infusion at rate 1000mg/hr
- Total: Total of all reporting groups
Arm/Group | Vancomycin Continous Infusion | Intermittent Infusion | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (14.1) | 53.7 (13.5) | 56.8 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 16 | 12 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved the Target Vancomycin Concentration
Description: The therapeutic level was defined as 15-20 mcg/mL for IIV and 15-25 mcg/mL for CIV
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin With Continuous Infusion | Vancomycin With Intermittent Dose Interval
Number analyzed (Participants) | 22 | 22
Participants | 20 | 5

2. Secondary Outcome: Time Required to Reach the Therapeutic Levels
Description: The therapeutic level was defined as 15-20 mcg/mL for IIV and 15-25 mcg/mL for CIV
Time Frame: as long as participants are receiving Vancomycin (mean (SD) 9 (3.8) days for continuous, 8.4 (4.1) days for intermittent)
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Vancomycin Continous Infusion: continuous 24 hours intravenous infusion
  Vancomycin continuous infusion: Vancomycin 24 hour intravenous continuous infusion
Arm/Group | Vancomycin Continous Infusion | Intermittent Infusion
Number analyzed (Participants) | 22 | 22
hours | 26.1 (7) | 54.1 (25.8)

3. Secondary Outcome: Vancomycin Concentration at 24 Hours
Description: The therapeutic level was defined as 15-20 mcg/mL for IIV and 15-25 mcg/mL for CIV
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Vancomycin Continous Infusion | Intermittent Infusion
Number analyzed (Participants) | 22 | 22
mcg/mL | 19.9 (3.7) | 14.2 (6.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while subjects are receiving vancomycin therapy.
Description: Nephrotoxicity was defined as an increase in serum creatinine (SCr) by 0.5 mg/dL or at least a 50% increase from baseline over 2 consecutive SCr values.
Arm/Group | Vancomycin Continous Infusion | Intermittent Infusion
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vancomycin Continous Infusion (N=22) | Intermittent Infusion (N=22)
Nephrotoxicity (Renal and urinary disorders) | 1 | 4 — Nephrotoxicity was defined as an increase in serum creatinine (SCr) by 0.5 mg/dL or at least a 50% increase from baseline over 2 consecutive SCr values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes